CLINICAL TRIAL: NCT04475393
Title: Multicentric Prospective Cohort Study in Patients With Irreversible Biventricular Heart Failure to Assess the Efficacy and Safety of Carmat TAH, Its Clinical Utility and Cost, as a Bridge to Transplantation
Brief Title: Carmat Total Artificial Heart as a Bridge to Transplant in Patients With Advanced Heart Failure
Acronym: EFICAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmat SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR2019-FR
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carmat TAH (Experimental): Subjects implanted with Carmat TAH
  Interventions: Device: Carmat Total Artificial Heart

INTERVENTIONS:
Device: Carmat Total Artificial Heart — Heart Replacement Therapy

SUMMARY:
The objective of this clinical investigation is to evaluate the efficacy and the safety of the Carmat Total Artificial Heart for the treatment of refractory advanced heart failure in transplant eligible patients.

DETAILED DESCRIPTION:
A selection committee (composed of two independent experts in the field of cardiovascular surgery/cardiology and of PIs) assess the subject eligibility based on clinical and anatomic criteria. Clinically eligible patients will be distributed into two cohorts depending on their anatomic compatibility with the device:

* cohort 1: patients that are anatomically compatible will receive the Carmat TAH ;
* cohort 2: patients that are not anatomically compatible will receive standard therapy

The efficacy and safety of the Carmat TAH will be assessed in cohort 1 and compared to a level of efficacy defined by the published data on the commercially available TAH; and adjusted for INTERMACS patient profile.

The clinical utility and the costs of Carmat TAH will be assessed by comparing the cohort of subject receiving the Carmat TAH to the cohort of patients treated by standard therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years or older
2. Patient in the waiting list for heart transplant or temporarily contraindicated for heart transplant
3. On inotropes or cardiac Index (CI) < 2.2 L/min/m2
4. On Optimal Medical Management as judged by the investigator based on current Heart Failure practice guidelines (ESC/HAS)
5. Eligible to biventricular Mechanical Circulatory Support according to one of the following category:

   1. Biventricular failure with at least two of the following hemodynamic/ echocardiographic measurements implying right heart failure:

      * RVEF ≤ 30% or FAC < 35%
      * RVSWI ≤ 0.25 mmHg*L/m2
      * TAPSE ≤ 14mm
      * RV-to-LV end-diastolic diameter ratio > 0.72
      * CVP > 15 mmHg or persistence of echographic and/or biological signs of hepatic congestion
      * CVP-to-PCWP ratio > 0.63
      * PAP index <2
      * Tricuspid insufficiency grade 4
   2. Treatment-refractory recurrent and sustained ventricular tachycardia or ventricular fibrillation in the presence of untreatable arrhythmogenic pathologic substrate.
   3. Heart failure due to restrictive or constrictive physiology (e.g., hypertrophic cardiomyopathy, cardiac amyloidosis / senile or other infiltrative heart disease)
6. Anatomic compatibility confirmed using 3D imaging (CT-scan) and by the screening committee (for Cohort 1).
7. Patient's affiliation to health care insurance
8. Patient has signed the informed consent.

Exclusion Criteria:

1. Absolute contra-indication for heart transplant
2. Existence of any ongoing non-temporary mechanical circulatory support
3. Existence of any ongoing peripheral mechanical circulatory support such as ECMO, Impella (all types), IABP with a support duration > 21 days
4. Patient intubated and unconscious; or intubated and not awake
5. Known intolerance to anticoagulant or antiplatelet therapies or known Heparin Induced Thrombocytopenia.
6. Coagulopathy defined by platelets < 100G/l or INR ≥ 1.5 not due to anticoagulant therapy.
7. Known thrombophilia (Antithrombin III, protein C or S deficiency) or any recurrent venous thromboembolic events requiring long term curative oral anticoagulation.
8. Cerebrovascular accident < 3 months or symptomatic (Rankin score >1; Glasgow score < 14) or a known > 80% carotid stenosis.
9. Known abdominal or thoracic aortic aneurysm > 5 cm that has not been treated.
10. Severe end-organ dysfunction as per the following criteria:

    1. Total bilirubin > 45 µmol/l (2.65 mg/dl) or cirrhosis evidenced by ultrasound, IRM and positive biopsy
    2. GFR < 30ml/min/1.73m2 (with no hemodialysis)
11. History of severe Chronic Obstructive Pulmonary Disease or severe restrictive lung disease with FEV1/FVC <0.7 and FEV1<50% predicted.
12. Recent active blood stream infection confirmed by a positive hemoculture within 48 hours.
13. Documented amyloid light-chain (AL amyloidosis).
14. Hemodynamically significant peripheral vascular disease assessed by clinical exam.
15. Illness, other than heart disease, that would limit survival to less than 2 years.
16. Irreversible cognitive dysfunction, psycho-cognitive disabilities, psycho-social issues or psychiatric disease, likely to impair compliance with the study protocol and TAH management that in the opinion of the investigator could interfere with the ability to manage the therapy (i.e. non-compliance to heart failure therapy, uncontrolled diabetes, mental health issue, etc.).
17. Pregnancy or breast feeding (woman in childbearing age will have to show negative pregnancy test).
18. Patient is currently enrolled or has participated in the last 30 days in another therapeutic or interventional clinical study that is likely to confound the study results or affect the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Survival free of disabling stroke at 180 days post-implant | 180 days
  Success is defined as survival free of disabling stroke (Modified Rankin score >3) at 180 days after Carmat TAH
  implantation or transplanted if before 180 days.

SECONDARY OUTCOMES:
Overall survival | 180 days - 1 year
  Survival post-implant; Survival post-transplantation (Kaplan-Meier)
General Health Status change | 180 days - 1 and 2 years
  Measured with the EuroQol EQ-5D-5L questionnaire, health-related quality of life consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (EQ-5D-5L). The responses record five levels of severity (1:no problems; 2:slight problems; 3:moderate problems 4:severe problems; 5:extreme problems) within a particular EQ-5D dimension.
Change in functional status measured by the Six Minutes Walk Test | 180 days - 1 and 2 years
  The 6-min walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Change in functional status | 180 days - 1 and 2 years
  New York Heart Association (NYHA) functional classification (regression scale I, II, III, IV)
Adverse Events | 180 days - 1 and 2 years
  Adverse Event Rates will be captured per the INTERMACS definitions
Hospital re-admissions rate | 180 days - 1 and 2 years
  Rate of unplanned re-admissions to the hospital
Healthcare costs | 180 days - 1 and 2 years
  The healthcare resources used to treat the patient during the two-year period, including those related to selection, those related to waiting for transplantation (whatever the therapeutic strategy), to transplantation, post-transplant management and any adverse event
Quality Adjusted Life Years | 180 days - 1 and 2 years
  The Quality Adjusted Life Years, evaluated during the two-year period, values the health outcomes in a single measure by combining both quality of life (evaluated by EuroQol EQ-5D-5L) and lenght of life.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Jansen, MD, Study Director — Carmat SAS
Locations (10):
- France (10):
  - Hôpital Louis Pradel, Bron
  - CHU Dijon, Dijon
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Centre Hospitalier Régional Universitaire, Lille
  - CHRU Montpellier, Montpellier
  - Hôpital Laennec, Nantes
  - Groupe Hospitalier Pitié-Salpêtrière,, Paris
  - Hôpital Européen George Pompidou, Paris
  - Hôpital Pontchaillou, Rennes
  - Nouvel Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No